CLINICAL TRIAL: NCT03327688
Title: Point-of-care Ultrasound in Finland
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ossi Hannula (Other)
Collaborators: University of Eastern Finland (Other)
Responsible Party: Sponsor-Investigator, Ossi Hannula, MD, emergency medicine resident, Kuopio University Hospital
Organization: Kuopio University Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: KUH507T027
Record Dates: First submitted 2017-10-23; First posted 2017-10-31 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Deep Vein Thrombosis; Abdominal Aortic Aneurism; Pneumothorax; Gallbladder Diseases; Hydronephrosis; Pregnancy, Ectopic; Ascites; Pleural Effusion; Pericardial Effusion
Keywords: Focus assesment with sonography for trauma; POCUS; LOS; Point-of-care ultrasound; length of stay; cost-minimization; primary health care; Ultrasound; Emergency department
MeSH Terms: conditions — Venous Thrombosis; Pneumothorax; Gallbladder Diseases; Hydronephrosis; Pregnancy, Ectopic; Ascites; Pleural Effusion; Pericardial Effusion; Emergencies

STUDY DESIGN:
Intervention Model Description: Part 1: All referrals to hospital due to a suspected DVT before intervention in year 2014, vs all referrals due to a suspected DVT after intervention in year 2017.
  Part 2: POCUS group vs radiologist group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- POCUS group (Active Comparator): Point-of-care ultrasound
  Interventions: Diagnostic Test: Point-of-care ultrasound
- Radiologist group (No Intervention): Traditional diagnostic way
- DVT POCUS group (Active Comparator): DVT group after POCUS education
  Interventions: Diagnostic Test: Point-of-care ultrasound
- DVT traditional group (No Intervention): DVT group traditional diagnostic way before educational intervention

INTERVENTIONS:
Diagnostic Test: Point-of-care ultrasound — Point-of-care ultrasound performed by an emergency physician
  Arms: DVT POCUS group; POCUS group

SUMMARY:
This study has two aims.

1. Deep venous thrombosis (DVT) is a common suspected medical condition. If it cannot be excluded clinically and using D-dimer, ultrasound examination is required. An option for traditional radiologist-performed ultrasound is a 2-point compression ultrasound (2-CUS). The safety of this technique is proven. However there does not exist any data on costs comparing traditional and 2-CUS pathways in primary health care. This study will evaluate the total cost of both pathways by conducting a cost-minimization analysis. It will also study the effect of a simple ultrasound education on the referrals to hospital due to suspected DVT.

   Hypothesis 1: Short education in ultrasound will reduce significantly referrals to hospital and save resources.
2. Length of stay (LOS) in emergency department (ED) is related to increased mortality, morbidity, prolonged hospital stay and probably patient satisfaction. LOS of patients with a point-of-care ultrasound (POCUS) performed by an emergency physician (EP) will be compared to those that have a radiology performed ultrasound examination. Further examination and accuracy of POCUS will be noted.

Hypothesis 2: POCUS can shorten LOS significantly in selected clinical conditions

DETAILED DESCRIPTION:
This study has two aims.

1. Deep venous thrombosis is a common suspected medical condition. If it cannot be excluded clinically and using D-dimer, ultrasound examination is required. An option for traditional radiologist-performed ultrasound is a 2-point compression ultrasound (2-CUS). The safety of this technique is proven. However there does not exist any data on costs comparing traditional and 2-CUS pathways in primary health care. This study will evaluate the total cost of both pathways by conducting a cost-minimization analysis. It will also study the effect of a simple ultrasound education on the referrals to hospital due to suspected DVT. T

   he study is performed in Saarikka Primary Care Public Utility, Saarijärvi, Finland. There are 15 general practitioners (GP) working. During year 2014, 2 of them were performing 2-CUS. 9 of the other GPs were trained during years 2015-2016 to perform a 2-CUS and hence 11 of 15 GPs are able to do 2-CUS in 2017.

   This is a register study. Referrals to hospital in 2014 (pre-training) and 2017 (post-training) are examined and the difference is assumed to be because of training and new pathway. Based on population the expected number of referrals due to a suspected DVT should be approximately 100 annually and the expected number after intervention is 30. According to power analysis a reduction from 100 to 76 is statistically significant (p<0.05).

   Hypothesis 1: Short education in ultrasound will reduce significantly referrals to hospital and save resources.
2. Length of stay (LOS) in emergency department (ED) is related to increased mortality, morbidity, prolonged hospital stay and probably patient satisfaction. LOS of patients with a point-of-care ultrasound (POCUS) performed by an emergency physician (EP) will be compared to those that have a radiology performed ultrasound examination.

This part started in Central Finland Central Hospital and Kuopio University Hospital 10/2017. Tampere university hospital will start at 5/2018.

An average LOS in Central Finland Central hospital ED is approximately 150 minutes. In a randomly selected monday in January, 2017, the average time from a referral to radiologist to a finished radiologist statement was 86 minutes. The times in Kuopio university hospital are much longer.

When an EP decides to perform a POCUS exam, they will recruit the patient in the study and fill a simple structured form. It is up to the EP treating the patient to decide if the patients needs POCUS. No additional examination because of this study is made on the patient.

The detailed time stamps for the patient to register in the ED, first doctor visit and finished from the doctor are retrieved from the files. In a follow-up of 6 months it is noted if the patient had a further examination by radiologist and if it was an ultrasound, CT, or some other examination. The results from POCUS will be compared to the radiologist examination, surgery or autopsy results where available and appropriate.

The control group is found from picture archive system (PACS) system with going through ultrasound examinations on the same days as POCUS examinations are made, with a referral question that a POCUS could answer, and referring unit being emergency department, and the same time points will be recorded.

There exists plenty of research on a focused ultrasound examination performed mostly by emergency physicians. In certain clinical questions such as abdominal aorta aneurysm or gallbladder stones, the accuracy of POCUS is excellent.

There also exists some research on POCUS effect on LOS compared to a standard ultrasound examination performed mostly by a radiologist. The reduction in LOS has been huge.

There is no data on regarding the Finnish health care system in this field. Also this study aims to evaluate multiple POCUS indications in a single real life setting which is not published before.

Hypothesis 2: POCUS can shorten LOS significantly in selected clinical conditions

Quality assurance plan: non-existent Data checks: non-existent Source data verification: EP filling the research form fills in only the finding in POCUS. It cannot reliably be verified in any way. All other data comes from medical records.

Data dictionary: Non-existent for now Standard operation procedures: Non-existent

Sample size assesment:

Part 1: a whole year prior and after intervention is evaluated. According to power analysis, change from 100 to 76 would be statistically significant. A reduction of 100 to 30 is expected.

Part 2: According to expected LOS reduction of at least 86 minutes, the study should need only approximately 10 patients + control group to show statistical significance. However a group of 400 patients will be recruited. The purpose of this is to be able to perform quality sub-group analysis based on indication of POCUS but also the experience level of EP performing the POCUS examination.

Plan for missing data: The study form in part 2 is the only reliable source for the POCUS results and if this is missing, the patient must be excluded. All other data is derived from the medical files statistics and should reliable.

Statistical analysis: A cost-minimization analysis will be performed in part 1. Other statistical analysis methods will be decided later.

ELIGIBILITY:
Inclusion Criteria:

* Emergency department patient
* A suspected medical condition, that can be confirmed or excluded by basic POCUS exam, including: free fluid in pleura, pericardium or intraperitoneal space, abdominal aorta aneurysm, gallbladder stones, urine retention, deep venous thrombosis in lower limb, pneumothorax, early pregnancy with non-specified location (confirming intrauterine pregnancy), hydronephrosis.
* Emergency medicine specialist or resident decides to perform a POCUS exam

Exclusion Criteria:

* age under 18
* not able to give informed consent in Finnish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Length of stay in emergency department | Duration of a single emergency department visit. Up to 48 hours.
  time between registration in emergency department and "finished from doctor" sign.

SECONDARY OUTCOMES:
Need for follow-up radiologist performed imaging | 6 months
  If radiologist performed ultrasound exam is required, is it performed the same day, during same hospital day or later by appointment. Does the POCUS examination lead to other imaging modality while skipping radiologist performed ultrasound exam.
Accuracy of POCUS exam findings | 6 months
  POCUS findings are compared to any follow-up imaging by radiologist, surgery results or autopsy results when possible

CONTACTS AND LOCATIONS:
Overall Officials: Harri Hyppölä, docent, Principal Investigator — Kuopio University Hospital
Locations (4):
- Finland (4):
  - Central Finland central hospital, Jyväskylä
  - Kuopio university hospital, Kuopio
  - Saarikka Primary Care Public Utility, Saarijärvi
  - Tampere university hospital, Tampere

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bernstein SL, Aronsky D, Duseja R, Epstein S, Handel D, Hwang U, McCarthy M, John McConnell K, Pines JM, Rathlev N, Schafermeyer R, Zwemer F, Schull M, Asplin BR; Society for Academic Emergency Medicine, Emergency Department Crowding Task Force. The effect of emergency department crowding on clinically oriented outcomes. Acad Emerg Med. 2009 Jan;16(1):1-10. doi: 10.1111/j.1553-2712.2008.00295.x. Epub 2008 Nov 8. PMID 19007346
- [Background] Ross M, Brown M, McLaughlin K, Atkinson P, Thompson J, Powelson S, Clark S, Lang E. Emergency physician-performed ultrasound to diagnose cholelithiasis: a systematic review. Acad Emerg Med. 2011 Mar;18(3):227-35. doi: 10.1111/j.1553-2712.2011.01012.x. PMID 21401784
- [Background] Rubano E, Mehta N, Caputo W, Paladino L, Sinert R. Systematic review: emergency department bedside ultrasonography for diagnosing suspected abdominal aortic aneurysm. Acad Emerg Med. 2013 Feb;20(2):128-38. doi: 10.1111/acem.12080. PMID 23406071
- [Background] Stein JC, Wang R, Adler N, Boscardin J, Jacoby VL, Won G, Goldstein R, Kohn MA. Emergency physician ultrasonography for evaluating patients at risk for ectopic pregnancy: a meta-analysis. Ann Emerg Med. 2010 Dec;56(6):674-83. doi: 10.1016/j.annemergmed.2010.06.563. Epub 2010 Sep 15. PMID 20828874
- [Background] Park YH, Jung RB, Lee YG, Hong CK, Ahn JH, Shin TY, Kim YS, Ha YR. Does the use of bedside ultrasonography reduce emergency department length of stay for patients with renal colic?: a pilot study. Clin Exp Emerg Med. 2016 Dec 30;3(4):197-203. doi: 10.15441/ceem.15.109. eCollection 2016 Dec. PMID 28168226
- [Background] Wilson SP, Connolly K, Lahham S, Subeh M, Fischetti C, Chiem A, Aspen A, Anderson C, Fox JC. Point-of-care ultrasound versus radiology department pelvic ultrasound on emergency department length of stay. World J Emerg Med. 2016;7(3):178-82. doi: 10.5847/wjem.j.1920-8642.2016.03.003. PMID 27547276
- [Background] Alrajab S, Youssef AM, Akkus NI, Caldito G. Pleural ultrasonography versus chest radiography for the diagnosis of pneumothorax: review of the literature and meta-analysis. Crit Care. 2013 Sep 23;17(5):R208. doi: 10.1186/cc13016. PMID 24060427
- [Background] Birdwell BG, Raskob GE, Whitsett TL, Durica SS, Comp PC, George JN, Tytle TL, McKee PA. The clinical validity of normal compression ultrasonography in outpatients suspected of having deep venous thrombosis. Ann Intern Med. 1998 Jan 1;128(1):1-7. doi: 10.7326/0003-4819-128-1-199801010-00001. PMID 9424975
- [Background] Ten Cate-Hoek AJ, Toll DB, Buller HR, Hoes AW, Moons KG, Oudega R, Stoffers HE, van der Velde EF, van Weert HC, Prins MH, Joore MA. Cost-effectiveness of ruling out deep venous thrombosis in primary care versus care as usual. J Thromb Haemost. 2009 Dec;7(12):2042-9. doi: 10.1111/j.1538-7836.2009.03627.x. Epub 2009 Sep 28. PMID 19793189